CLINICAL TRIAL: NCT01014832
Title: An Efficacy and Safety Evaluation of Frequently Modified Intensive Insulin Therapy in Subjects With Uncontrolled Type-I or Type-2 Diabetes
Brief Title: Efficacy and Safety of Frequently Modified Intensive Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hygieia, Inc (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Israel Hodish MD. PhD., Hygieia INC.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hygieia study -2; CS950308 (Other: Hygieia INC.)
Record Dates: First submitted 2009-11-13; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes
Keywords: Diabetes, insulin.
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uncontrolled diabetes (Experimental): Uncontrolled diabetes
  Interventions: Drug: Intensive insulin therapy

INTERVENTIONS:
Drug: Intensive insulin therapy — Intensive insulin therapy
  Other Names: Basal-bolus insulin therapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of frequently modified intensive insulin therapy in patients with Type-2 and Type-1 diabetes mellitus.

DETAILED DESCRIPTION:
Insulin treatment is the mainstay of Type-1 diabetic management and one of the cornerstones in Type-2 diabetes. This treatment is based on multiple daily injections of different types of insulin. Patients follow their endocrinologists' directions by adhering to a set of recommended dosages and formulas, calculated by repeated blood glucose measurements. In order to maintain effective and safe management, glucose measurements are taken before meals and at bedtime, albeit imposing a heavy financial burden on a patient and their support system. For illustration, each disposable glucosemeter strip costs more than a dollar and needs to be replaced routinely 4 times daily, yielding an annual cost of more than $1500 per patient. Insulin dosages necessitate repeated adjustments to meet the patient's changing needs. Variations in food intake, body weight, physical activity, on going medical conditions and mood can impact a patient's insulin needs.

Accordingly, at each diabetic clinic appointment, the endocrinologist reviews the patient's glucose measurements and insulin doses to determine whether the insulin dosage needs to be adjusted. Unfortunately, limited appointment availability restricts insulin dosages adjustments to once every several months. Furthermore, as a result of the limited time allotted for each patient, new dosing recommendations are based on a review of only the most recent measurements. This drawback may be one of the chief causes of suboptimal management, with merely 38% of diabetic patients able to achieve proper control and mitigate detrimental complications.

Since the discovery of insulin by Frederick Grant Banting in 1921, only stringent glucose control by a regimen of multiple insulin injections has prevented microvascular and macrovascular complications in Type 1 diabetic patients. Moreover, insulin treatment amongst other treatment modalities has been shown to prevent microvascular and macrovascular complications in Type-2 diabetic patients. Incidentally, as the Type-2 diabetic epidemic expands, insulin treatment is becoming one of the main treatment modalities. Not taking into consideration availability, it has been established that more frequent patient-clinic interactions improve diabetic management in both Type-1 and Type-2 patients.

In a typical 3-6 month interval appointment, the endocrinologist would measure a patient's hemoglobin A1c (HbA1c) to determine the quality of the last 3 months control. This value, is linearly correlated to mean glucose levels at that 3 months period and, therefore, can be predicted according to the measurements. We used anonymous records of glucose measurements to perform preliminary statistical analysis. Our results indicate that a patient's glucose level is a highly non-stationary process, with strong variations in both mean and standard deviation (SD) from one week to another. In many patients with excessive HbA1c, which are at levels that diabetic complications are likely to ensue, the endocrinologist is obligated to adjust the insulin dosage based on a review of the patient's most recent glucose values and the values of the past several weeks. Furthermore, since appointment timing is random and independent from the patient's measurements, random trends in glucose values may be identified that lead to different conclusions. For illustration, if a patient's appointment happens to occur when his glucose values randomly trend up, the endocrinologist may choose to increase insulin doses. On the other hand, if the appointment occurs at a time when the glucose levels trend down, he may act oppositely. The required frequency of follow-up and dose adjustment that yields better patient control is yet to be determined.

Studies have shown that case management in patients with Type-2 diabetes can allow better control of HbA1c levels. These studies have involved using qualified medical professionals (ie, nurses, pharmacists, physician's assistants) as intervention methods, as well as providing counseling and follow-up calls to help patients with improved self-management of diabetes.

This study is designed to show that weekly insulin dosage adjustments for intensive insulin therapy are superior to conservative, infrequent adjustments during clinical appointments in both Type-1 and Type-2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for inclusion in the study are those who:

1. are male or female, 25 to 65 years of age;
2. are of any ethnic background;
3. meet the criteria for either population I or population II;
4. if a female of child-bearing potential will submit to a urine pregnancy test (UPT) at Visit 1;
5. can provide their previous 12 months of lab results (at least one set of blood count, kidney functions, and liver enzymes); and
6. read, understand, and sign an informed consent document which contains a Health Information Portability and Accountability Act (HIPAA) authorization after being advised of the nature of the study.

Population I inclusion criteria:

Individuals eligible for inclusion in population I are those who:

1. meet the standard criteria for enrollment in the study;
2. have been clinically diagnosed compatible with Type-2 diabetes for at least 1 year;
3. take insulin injections for the past 6 months;
4. have or have not been using an oral agent within the past 6 months;
5. have sufficient medical insurance coverage to cover intensive insulin therapy including Lantus® and Humalog®/Novolog® as well as test-strips cost for testing their blood glucose levels at least 4 times per day;
6. are willing to stop anti-diabetic agents (except Metformin);
7. are willing to accept intensive insulin therapy with at least 4 daily insulin injections;
8. consistently record their glucose measurements and insulin doses in a log book and have their previous readings ready for review; and
9. have a Hemoglobin-A1c (HbA1c) of 7.6% or greater, to be drawn at Visit 1.

Population II inclusion criteria:

Individuals eligible for inclusion in population II are those who:

1. meet the standard criteria for enrollment in the study;
2. have been clinically diagnosed compatible with Type-1 diabetes for at least 1 year;
3. treated with both long acting insulin analog (ie, Insulin Glargine) and short acting insulin analog (ie, Insulin Lispro or Insulin Aspart) with a total daily insulin dose of 25 units or more
4. are currently using carbohydrate counting in their regimen or have been trained to employ this technique during the last 2 years;
5. consistently record their glucose measurements and insulin doses in a log book and have their previous readings for review; and
6. have a HbA1c of 7.6% or greater, to be drawn at Visit 1.

Exclusion Criteria:

Individuals excluded from participation in the study are those who:

1. have a history of greater than 2 episodes of severe hypoglycemia (See Section 5.4) in the past year or hypoglycemic unawareness;
2. have a significant physical, psychological, or cognitive impairment that would prohibit adherence to an intensive insulin therapy program;
3. have any severe cardiovascular disease including a history of congestive heart failure (New York Heart Association [NYHA] 3 or 4), unstable angina, myocardial infarction or stroke that occurred within 6 months prior to enrollment
4. have a history of severe anemia with a hematocrit less than 25% in women or 30% in men;
5. have a history of renal disease (ie, serum creatinine level greater than 2.0 mg/dl);
6. have a history of active cancer or cancer in the past 2 years (except non-melanoma skin cancer);
7. are receiving chemotherapy or radiation therapy;
8. have a history of significant liver disease including cirrhosis or elevated liver function tests (AST and ALT) greater than 3 times the upper limit of normal values;
9. have a body mass index (BMI) greater than 45 kg/m2; and/or
10. are pregnant, plan to become pregnant during the study period, or are breastfeeding.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | 12 weeks
Mean weekly glucose | 12 weeks
Frequency of hypoglycemia | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Israel Hodish, MD. PhD., Study Director — Hygieia, Inc; Michael Casser, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research INC., Paramus, New Jersey, United States